CLINICAL TRIAL: NCT03012984
Title: Impact of Dexmedetomidine Supplemented Analgesia on Incidence of Delirium in Elderly Patients After Cancer Surgery: a Multicenter Randomized Controlled Trial
Brief Title: Dexmedetomidine Supplemented Analgesia and Incidence of Postoperative Delirium
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Peking University First Hospital (Other)
Collaborators: Affiliated Hospital of Hebei University (Other); Qingdao Municipal Hospital (Other); The Second Affiliated Hospital of Air Force Medical University (Unknown); Peking University International Hospital (Other); Guizhou Provincial People's Hospital (Other); The Third Xiangya Hospital of Central South University (Other); Shanxi Provincial Cancer Hospital (Unknown); Tianjin Hospital of ITCWM-Nankai Hospital (Unknown); Chongqing University Fuling Hospital (Unknown); The Third Central Hospital of Tianjin (Unknown); Xiyuan Hospital of China Academy of Chinese Medical Sciences (Other)
Responsible Party: Principal Investigator, Dong-Xin Wang, Professor and Chairman, Department of Anesthesiology, Peking University First Hospital
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 2016-10
Record Dates: First submitted 2016-12-31; First posted 2017-01-06 (Estimated); Last update posted 2026-01-08 (Actual); Status verified 2026-01

CONDITIONS: Elderly; Surgery; Analgesia; Dexmedetomidine; Complication, Postoperative; Delirium
Keywords: elderly; surgery; analgesia; dexmedetomidine; delirium
MeSH Terms: conditions — Agnosia; Postoperative Complications; Delirium

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Dexmedetomidine group (Experimental): Dexmedetomidine supplemented morphine analgesia will be provided for patients in this group in the form of patient-controlled intravenous analgesia. The formula contains a mixture of morphine (0.5 mg/ml) and dexmedetomidine (1.25 ug/ml), diluted with normal saline to a total volume of 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time from 6 to 8 minutes.
  Interventions: Drug: Dexmedetomidine supplemented morphine analgesia
- Control group (Placebo Comparator): Morphine analgesia will be provided for patients in this group in the form of patient-controlled intravenous analgesia. The formula contains morphine (0.5 mg/ml), diluted with normal saline to a total volume of 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with patient-controlled bolus of 2 ml each time and a lockout time from 6 to 8 minutes.
  Interventions: Drug: Morphine analgesia

INTERVENTIONS:
Drug: Dexmedetomidine supplemented morphine analgesia — Patients in this group will receive patient-controlled intravenous analgesia for 3 days after surgery. The formula is a mixture of dexmedetomidine (1.25 ug/ml) and morphine (0.5 mg/ml), diluted with normal saline to 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml each time and a lockout time from 6 to 8 minutes according to patients' condition.
  Arms: Dexmedetomidine group
Drug: Morphine analgesia — Patients in this group will receive patient-controlled intravenous analgesia for 3 days after surgery. The formula is morphine (0.5 mg/ml) diluted with normal saline to 160 ml. 5-HT3 receptor antagonist is added when necessary. The analgesic pump is set to administer a background infusion at a rate of 1 ml/h, with a bolus dose of 2 ml each time and a lockout time from 6 to 8 minutes according to patients' condition.
  Arms: Control group

SUMMARY:
Delirium is a frequently occurred cerebral complication in elderly patients after surgery, and its occurrence is associated with worse outcomes. Sleep disturbances is considered to be one of the most important risk factors of postoperative delirium. Previous studies showed that, for elderly patients admitted to the ICU after surgery, low-dose dexmedetomidine infusion improved the quality of sleep and decreased the incidence of delirium. The investigators hypothesize that, for elderly patients after cancer surgery, dexmedetomidine supplemented analgesia can also decrease the incidence of delirium, possibly by improving sleep quality. The purpose of this multicenter, randomized controlled trial is to investigate the impact of dexmedetomidine supplemented analgesia on the incidence of delirium in elderly patients after cancer surgery.

DETAILED DESCRIPTION:
Delirium is a state of acutely occurred and transient cerebral dysfunction. It is a common complication in elderly patients after surgery. A systematic review showed that an average of 36.8% (range 0 to 73.5%) of surgical patients developed postoperative delirium, and its occurrence increased with age. According to our previous studies, postoperative delirium developed in 51.0% of patients after cardiac surgery and in 44.5% of patients after non-cardiac surgery. The occurrence of delirium is associated with worse short-term outcomes, including increased postoperative complications, prolonged hospital stay, and increased in-hospital mortality; it is also associated with worse longterm outcomes, including declined cognitive function, decreased quality of life, and increased post-hospital mortality. Delirium is the result of multiple factors. Studies showed that postoperative pain is an important risk factor of delirium, whereas good postoperative analgesia reduces the incidence of delirium. For postoperative patients, sleep disturbances occurs frequently and increases the risk of delirium, whereas improving sleep quality reduces the incidence of delirium. Furthermore, the studies found that surgery related inflammatory response also plays an important role in the development of delirium.

Dexmedetomidine is a highly selective alpha-2 (α2) adrenoreceptor agonist that provides anxiolysis, sedation, hypnosis and analgesia. It exerts the sedative and hypnotic effects by activating the endogenous sleep pathways, and produces a condition similar to phase 2 non-rapid eye movement sleep. For patients undergoing mechanical ventilation in the ICU, dexmedetomidine sedation helps to maintain a normal circadian rhythm of sleep and improves sleep architecture. Dexmedetomidine also provides analgesic effect by activating α2 adrenergic receptors in the dorsal horn of spinal cord. When used as a supplemental drug it decreases intraoperative and postoperative requirement of opioids. Moreover, animal studies showed that dexmedetomidine significantly inhibits the degree of inflammatory response induced by endotoxin or during spinal cord injury. In clinical studies, dexmedetomidine attenuates the degree of inflammatory response following Coronary Artery Bypass Grafting surgery.

These effects of dexmedetomidine make it suitable for prevention of postoperative delirium in high-risk patients. Studies have shown that, for ICU patients requiring mechanical ventilation, sedation with dexmedetomidine reduces the incidence of delirium when compared with other sedatives; for postoperative patients, dexmedetomidine administered in combined with opioids improves analgesia and reduces opioid requirements. A recent study showed that, for elderly patients admitted to the ICU after surgery, low-dose dexmedetomidine infusion (at a rate of 0.1 ug/kg/h, for an average of 15 hours) improves analgesia for up to 24 hours, ameliorates subjective sleep quality for up to 3 days, and reduces the incidence of delirium during the first 7 postoperative days. The investigators hypothesized that the use of dexmedetomidine as a supplement to patient-controlled intravenous analgesia may also reduce the incidence of postoperative delirium.

ELIGIBILITY:
Inclusion Criteria:

* Age >= 65 years, < 90 years;
* Scheduled to undergo curative resection for primary solid organ cancer under general anesthesia, with an expected duration of surgery >=2 hours;
* Planned to use patient-controlled intravenous analgesia after surgery;
* Provide written informed consent.

Exclusion Criteria:

* Preoperative history of schizophrenia, epilepsy, parkinsonism or myasthenia gravis;
* Preoperative radio- or chemotherapy;
* Inability to communicate in the preoperative period because of coma, profound dementia or language barrier;
* Preoperative obstructive sleep apnea (previously diagnosed as obstructive sleep apnea, or a STOP-Bang score >= 3 and serum HCO3- >= 28 mmol/L);
* Brain trauma or neurosurgery;
* Preoperative left ventricular ejection fraction < 30%, sick sinus syndrome, severe sinus bradycardia (< 50 beats per minute), or second-degree or above atrioventricular block without pacemaker;
* Severe hepatic dysfunction (Child-Pugh class C) or severe renal dysfunction (requirement of renal replacement therapy before surgery);
* ASA classification >= IV.

Ages: 65 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 1500 (Actual)
Dates: Start 2017-01-06 (Actual); Primary Completion 2022-05-12 (Actual); Study Completion 2022-06-11 (Actual)

PRIMARY OUTCOMES:
Incidence of delirium within 5 days after surgery | During the first 5 days after surgery
  Incidence of delirium within 5 days after surgery

SECONDARY OUTCOMES:
Daily prevalence of delirium during the first 5 postoperative days | During the first 5 postoperative days
  Daily prevalence of delirium during the first 5 postoperative days
Length of stay in hospital after surgery | Up to 30 days after surgery
  Length of stay in hospital after surgery
Incidence of non-delirium complications after surgery | Up to 30 days after surgery
  Incidence of non-delirium complications after surgery
30-day all-cause mortality after surgery | At the time of 30 days after surgery
  30-day all-cause mortality after surgery
Quality of life in survival patients on the 30th day after surgery | On the 30th day after surgery
  Assessed with World Health Organization Quality of Life-Bref (WHOQOL-BREF)
Cognitive function in survival patients on the 30th day after surgery | On the 30th day after surgery
  Assessed with Telephone Interview for Cognitive Status-Modified (TICS-M)

OTHER OUTCOMES:
Richmond Agitation-Sedation Scale (RASS) score during the first 5 days after surgery | During the first 5 days after surgery
  Richmond Agitation-Sedation Scale (RASS) score during the first 5 days after surgery
Cumulative morphine consumption during the first 3 days after surgery | During the first 3 days after surgery
  Cumulative morphine consumption during the first 3 days after surgery
Numeric Rating Scale (NRS) pain score during the first 5 days after surgery | During the first 5 days after surgery
  Numeric Rating Scale (NRS) pain score during the first 5 days after surgery
Numeric Rating Scale (NRS) sleep quality score during the first 5 days after surgery | During the first 5 days after surgery
  Numeric Rating Scale (NRS) sleep quality score during the first 5 days after surgery

CONTACTS AND LOCATIONS:
Overall Officials: Dong-Xin Wang, MD,PhD, Principal Investigator — Peking University First Hospital
Locations (12):
- China (12):
  - Peking University First Hospital, Beijing, Beijing Municipality
  - Xiyuan Hospital of China Academy of Chinese Medical Sciences, Beijing, Beijing Municipality
  - Peking University International Hospital, Beijing, Beijing Municipality
  - Chongqing University Fuling Hospital, Chongqing, Chongqing Municipality
  - Guizhou Provincial People's Hospital, Guiyang, Guizhou
  - Affiliated Hospital of Hebei University, Baoding, Hebei
  - The Third Xiangya Hospital of Central South University, Changsha, Hunan
  - The Second Affiliated Hospital of Air Force Medical University, Xi'an, Shaanxi
  - Qingdao Municipal Hospital, Qingdao, Shandong
  - Shanxi Provincial Cancer Hospital, Taiyuan, Shanxi
  - Tianjin Hospital of ITCWM-Nankai Hospital, Tianjin, Tianjin Municipality
  - The Third Central Hospital of Tianjin, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Friese RS. Sleep and recovery from critical illness and injury: a review of theory, current practice, and future directions. Crit Care Med. 2008 Mar;36(3):697-705. doi: 10.1097/CCM.0B013E3181643F29. PMID 18176314
- [Background] Ma J, Zhang XL, Wang CY, Lin Z, Tao JR, Liu HC. Dexmedetomidine alleviates the spinal cord ischemia-reperfusion injury through blocking mast cell degranulation. Int J Clin Exp Med. 2015 Sep 15;8(9):14741-9. eCollection 2015. PMID 26628956
- [Background] Bekker A, Haile M, Kline R, Didehvar S, Babu R, Martiniuk F, Urban M. The effect of intraoperative infusion of dexmedetomidine on the quality of recovery after major spinal surgery. J Neurosurg Anesthesiol. 2013 Jan;25(1):16-24. doi: 10.1097/ANA.0b013e31826318af. PMID 22824921
- [Background] Mu DL, Wang DX, Li LH, Shan GJ, Li J, Yu QJ, Shi CX. High serum cortisol level is associated with increased risk of delirium after coronary artery bypass graft surgery: a prospective cohort study. Crit Care. 2010;14(6):R238. doi: 10.1186/cc9393. Epub 2010 Dec 30. PMID 21192800
- [Background] Dyer CB, Ashton CM, Teasdale TA. Postoperative delirium. A review of 80 primary data-collection studies. Arch Intern Med. 1995 Mar 13;155(5):461-5. doi: 10.1001/archinte.155.5.461. PMID 7864702
- [Background] McDaniel M, Brudney C. Postoperative delirium: etiology and management. Curr Opin Crit Care. 2012 Aug;18(4):372-6. doi: 10.1097/MCC.0b013e3283557211. PMID 22732435
- [Background] Shi CM, Wang DX, Chen KS, Gu XE. Incidence and risk factors of delirium in critically ill patients after non-cardiac surgery. Chin Med J (Engl). 2010 Apr 20;123(8):993-9. PMID 20497703
- [Background] Lat I, McMillian W, Taylor S, Janzen JM, Papadopoulos S, Korth L, Ehtisham A, Nold J, Agarwal S, Azocar R, Burke P. The impact of delirium on clinical outcomes in mechanically ventilated surgical and trauma patients. Crit Care Med. 2009 Jun;37(6):1898-905. doi: 10.1097/CCM.0b013e31819ffe38. PMID 19384221
- [Background] Quinlan N, Rudolph JL. Postoperative delirium and functional decline after noncardiac surgery. J Am Geriatr Soc. 2011 Nov;59 Suppl 2:S301-4. doi: 10.1111/j.1532-5415.2011.03679.x. PMID 22091577
- [Background] Lescot T, Karvellas CJ, Chaudhury P, Tchervenkov J, Paraskevas S, Barkun J, Metrakos P, Goldberg P, Magder S. Postoperative delirium in the intensive care unit predicts worse outcomes in liver transplant recipients. Can J Gastroenterol. 2013 Apr;27(4):207-12. doi: 10.1155/2013/289185. PMID 23616958
- [Background] Abelha FJ, Luis C, Veiga D, Parente D, Fernandes V, Santos P, Botelho M, Santos A, Santos C. Outcome and quality of life in patients with postoperative delirium during an ICU stay following major surgery. Crit Care. 2013 Oct 29;17(5):R257. doi: 10.1186/cc13084. PMID 24168808
- [Background] Pisani MA, Kong SY, Kasl SV, Murphy TE, Araujo KL, Van Ness PH. Days of delirium are associated with 1-year mortality in an older intensive care unit population. Am J Respir Crit Care Med. 2009 Dec 1;180(11):1092-7. doi: 10.1164/rccm.200904-0537OC. Epub 2009 Sep 10. PMID 19745202
- [Background] Bickel H, Gradinger R, Kochs E, Forstl H. High risk of cognitive and functional decline after postoperative delirium. A three-year prospective study. Dement Geriatr Cogn Disord. 2008;26(1):26-31. doi: 10.1159/000140804. Epub 2008 Jun 24. PMID 18577850
- [Background] Van Rompaey B, Schuurmans MJ, Shortridge-Baggett LM, Truijen S, Elseviers M, Bossaert L. Long term outcome after delirium in the intensive care unit. J Clin Nurs. 2009 Dec;18(23):3349-57. doi: 10.1111/j.1365-2702.2009.02933.x. Epub 2009 Sep 4. PMID 19735334
- [Background] Ouimet S, Kavanagh BP, Gottfried SB, Skrobik Y. Incidence, risk factors and consequences of ICU delirium. Intensive Care Med. 2007 Jan;33(1):66-73. doi: 10.1007/s00134-006-0399-8. Epub 2006 Nov 11. PMID 17102966
- [Background] Stuck A, Clark MJ, Connelly CD. Preventing intensive care unit delirium: a patient-centered approach to reducing sleep disruption. Dimens Crit Care Nurs. 2011 Nov-Dec;30(6):315-20. doi: 10.1097/DCC.0b013e31822fa97c. PMID 21983504
- [Background] Siddiqi N, Harrison JK, Clegg A, Teale EA, Young J, Taylor J, Simpkins SA. Interventions for preventing delirium in hospitalised non-ICU patients. Cochrane Database Syst Rev. 2016 Mar 11;3(3):CD005563. doi: 10.1002/14651858.CD005563.pub3. PMID 26967259
- [Background] Kosar CM, Tabloski PA, Travison TG, Jones RN, Schmitt EM, Puelle MR, Inloes JB, Saczynski JS, Marcantonio ER, Meagher D, Reid MC, Inouye SK. EFFECT OF PREOPERATIVE PAIN AND DEPRESSIVE SYMPTOMS ON THE DEVELOPMENT OF POSTOPERATIVE DELIRIUM. Lancet Psychiatry. 2014 Nov;1(6):431-436. doi: 10.1016/S2215-0366(14)00006-6. PMID 25642413
- [Background] Halaszynski TM. Pain management in the elderly and cognitively impaired patient: the role of regional anesthesia and analgesia. Curr Opin Anaesthesiol. 2009 Oct;22(5):594-9. doi: 10.1097/ACO.0b013e32833020dc. PMID 19623056
- [Background] Rudolph JL, Ramlawi B, Kuchel GA, McElhaney JE, Xie D, Sellke FW, Khabbaz K, Levkoff SE, Marcantonio ER. Chemokines are associated with delirium after cardiac surgery. J Gerontol A Biol Sci Med Sci. 2008 Feb;63(2):184-9. doi: 10.1093/gerona/63.2.184. PMID 18314455
- [Background] Brummel NE, Girard TD. Preventing delirium in the intensive care unit. Crit Care Clin. 2013 Jan;29(1):51-65. doi: 10.1016/j.ccc.2012.10.007. PMID 23182527
- [Background] de Rooij SE, van Munster BC, Korevaar JC, Levi M. Cytokines and acute phase response in delirium. J Psychosom Res. 2007 May;62(5):521-5. doi: 10.1016/j.jpsychores.2006.11.013. PMID 17467406
- [Background] Mo Y, Zimmermann AE. Role of dexmedetomidine for the prevention and treatment of delirium in intensive care unit patients. Ann Pharmacother. 2013 Jun;47(6):869-76. doi: 10.1345/aph.1AR708. PMID 23719785
- [Background] Huupponen E, Maksimow A, Lapinlampi P, Sarkela M, Saastamoinen A, Snapir A, Scheinin H, Scheinin M, Merilainen P, Himanen SL, Jaaskelainen S. Electroencephalogram spindle activity during dexmedetomidine sedation and physiological sleep. Acta Anaesthesiol Scand. 2008 Feb;52(2):289-94. doi: 10.1111/j.1399-6576.2007.01537.x. Epub 2007 Nov 14. PMID 18005372
- [Background] Oto J, Yamamoto K, Koike S, Onodera M, Imanaka H, Nishimura M. Sleep quality of mechanically ventilated patients sedated with dexmedetomidine. Intensive Care Med. 2012 Dec;38(12):1982-9. doi: 10.1007/s00134-012-2685-y. Epub 2012 Sep 8. PMID 22961436
- [Background] Coull JT, Jones ME, Egan TD, Frith CD, Maze M. Attentional effects of noradrenaline vary with arousal level: selective activation of thalamic pulvinar in humans. Neuroimage. 2004 May;22(1):315-22. doi: 10.1016/j.neuroimage.2003.12.022. PMID 15110021
- [Background] Memis D, Hekimoglu S, Vatan I, Yandim T, Yuksel M, Sut N. Effects of midazolam and dexmedetomidine on inflammatory responses and gastric intramucosal pH to sepsis, in critically ill patients. Br J Anaesth. 2007 Apr;98(4):550-2. doi: 10.1093/bja/aem017. No abstract available. PMID 17363413
- [Background] Tasdogan M, Memis D, Sut N, Yuksel M. Results of a pilot study on the effects of propofol and dexmedetomidine on inflammatory responses and intraabdominal pressure in severe sepsis. J Clin Anesth. 2009 Sep;21(6):394-400. doi: 10.1016/j.jclinane.2008.10.010. PMID 19833271
- [Background] Stone LS, MacMillan LB, Kitto KF, Limbird LE, Wilcox GL. The alpha2a adrenergic receptor subtype mediates spinal analgesia evoked by alpha2 agonists and is necessary for spinal adrenergic-opioid synergy. J Neurosci. 1997 Sep 15;17(18):7157-65. doi: 10.1523/JNEUROSCI.17-18-07157.1997. PMID 9278550
- [Background] Szumita PM, Baroletti SA, Anger KE, Wechsler ME. Sedation and analgesia in the intensive care unit: evaluating the role of dexmedetomidine. Am J Health Syst Pharm. 2007 Jan 1;64(1):37-44. doi: 10.2146/ajhp050508. PMID 17189578
- [Background] Arcangeli A, D'Alo C, Gaspari R. Dexmedetomidine use in general anaesthesia. Curr Drug Targets. 2009 Aug;10(8):687-95. doi: 10.2174/138945009788982423. PMID 19702517
- [Background] Taniguchi T, Kidani Y, Kanakura H, Takemoto Y, Yamamoto K. Effects of dexmedetomidine on mortality rate and inflammatory responses to endotoxin-induced shock in rats. Crit Care Med. 2004 Jun;32(6):1322-6. doi: 10.1097/01.ccm.0000128579.84228.2a. PMID 15187514
- [Background] Can M, Gul S, Bektas S, Hanci V, Acikgoz S. Effects of dexmedetomidine or methylprednisolone on inflammatory responses in spinal cord injury. Acta Anaesthesiol Scand. 2009 Sep;53(8):1068-72. doi: 10.1111/j.1399-6576.2009.02019.x. Epub 2009 Jun 10. PMID 19519725
- [Background] Ueki M, Kawasaki T, Habe K, Hamada K, Kawasaki C, Sata T. The effects of dexmedetomidine on inflammatory mediators after cardiopulmonary bypass. Anaesthesia. 2014 Jul;69(7):693-700. doi: 10.1111/anae.12636. Epub 2014 Apr 28. PMID 24773263
- [Background] Pandharipande PP, Pun BT, Herr DL, Maze M, Girard TD, Miller RR, Shintani AK, Thompson JL, Jackson JC, Deppen SA, Stiles RA, Dittus RS, Bernard GR, Ely EW. Effect of sedation with dexmedetomidine vs lorazepam on acute brain dysfunction in mechanically ventilated patients: the MENDS randomized controlled trial. JAMA. 2007 Dec 12;298(22):2644-53. doi: 10.1001/jama.298.22.2644. PMID 18073360
- [Background] Riker RR, Shehabi Y, Bokesch PM, Ceraso D, Wisemandle W, Koura F, Whitten P, Margolis BD, Byrne DW, Ely EW, Rocha MG; SEDCOM (Safety and Efficacy of Dexmedetomidine Compared With Midazolam) Study Group. Dexmedetomidine vs midazolam for sedation of critically ill patients: a randomized trial. JAMA. 2009 Feb 4;301(5):489-99. doi: 10.1001/jama.2009.56. Epub 2009 Feb 2. PMID 19188334
- [Background] Peng K, Liu HY, Wu SR, Cheng H, Ji FH. Effects of Combining Dexmedetomidine and Opioids for Postoperative Intravenous Patient-controlled Analgesia: A Systematic Review and Meta-analysis. Clin J Pain. 2015 Dec;31(12):1097-104. doi: 10.1097/AJP.0000000000000219. PMID 25654534
- [Background] Su X, Meng ZT, Wu XH, Cui F, Li HL, Wang DX, Zhu X, Zhu SN, Maze M, Ma D. Dexmedetomidine for prevention of delirium in elderly patients after non-cardiac surgery: a randomised, double-blind, placebo-controlled trial. Lancet. 2016 Oct 15;388(10054):1893-1902. doi: 10.1016/S0140-6736(16)30580-3. Epub 2016 Aug 16. PMID 27542303
- [Background] Hofer SO, Molema G, Hermens RA, Wanebo HJ, Reichner JS, Hoekstra HJ. The effect of surgical wounding on tumour development. Eur J Surg Oncol. 1999 Jun;25(3):231-43. doi: 10.1053/ejso.1998.0634. PMID 10336800
- [Background] Nguyen DP, Li J, Tewari AK. Inflammation and prostate cancer: the role of interleukin 6 (IL-6). BJU Int. 2014 Jun;113(6):986-92. doi: 10.1111/bju.12452. PMID 24053309
- [Background] Schrepf A, Thaker PH, Goodheart MJ, Bender D, Slavich GM, Dahmoush L, Penedo F, DeGeest K, Mendez L, Lubaroff DM, Cole SW, Sood AK, Lutgendorf SK. Diurnal cortisol and survival in epithelial ovarian cancer. Psychoneuroendocrinology. 2015 Mar;53:256-67. doi: 10.1016/j.psyneuen.2015.01.010. Epub 2015 Jan 20. PMID 25647344
- [Background] Roy S, Ninkovic J, Banerjee S, Charboneau RG, Das S, Dutta R, Kirchner VA, Koodie L, Ma J, Meng J, Barke RA. Opioid drug abuse and modulation of immune function: consequences in the susceptibility to opportunistic infections. J Neuroimmune Pharmacol. 2011 Dec;6(4):442-65. doi: 10.1007/s11481-011-9292-5. Epub 2011 Jul 26. PMID 21789507
- [Background] Vassou D, Notas G, Hatzoglou A, Castanas E, Kampa M. Opioids increase bladder cancer cell migration via bradykinin B2 receptors. Int J Oncol. 2011 Sep;39(3):697-707. doi: 10.3892/ijo.2011.1063. Epub 2011 Jun 3. PMID 21643624
- [Background] Fujioka N, Nguyen J, Chen C, Li Y, Pasrija T, Niehans G, Johnson KN, Gupta V, Kratzke RA, Gupta K. Morphine-induced epidermal growth factor pathway activation in non-small cell lung cancer. Anesth Analg. 2011 Dec;113(6):1353-64. doi: 10.1213/ANE.0b013e318232b35a. Epub 2011 Oct 14. PMID 22003224
- [Background] Alexopoulou C, Kondili E, Diamantaki E, Psarologakis C, Kokkini S, Bolaki M, Georgopoulos D. Effects of dexmedetomidine on sleep quality in critically ill patients: a pilot study. Anesthesiology. 2014 Oct;121(4):801-7. doi: 10.1097/ALN.0000000000000361. PMID 24988068